CLINICAL TRIAL: NCT04005625
Title: Features of Microcrystalline Polyarthritis Treated by Biologics and Evolution - FUMBLE Study
Brief Title: Biotherapy Treatment on Features of Microcrystalline Polyarthritis
Acronym: FUMBLE
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC19.0056
Record Dates: First submitted 2019-03-29; First posted 2019-07-02 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Crystal-Induced Arthritis
Keywords: Crystal-Induced Arthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study will involve adult patient who had received any biologic agent for microcrystalline disease in western France (Tours, Le Mans, Orléans, Angers, Rennes, Poitiers et Brest) between 01/01/2010 and 31/12/2018.

Investigators will answer retrospectively a questionnaire that covers patient and disease data, biologic agent use, efficacy and adverse events.

DETAILED DESCRIPTION:
This is a retrospective multicentric study of all patients treated by biologic for microcrystalline disease in France in western France (Tours, Le Mans, Nantes, La Roche sur Yon, Orléans, Angers, Rennes, Poitiers et Brest) between 01/01/2010 and 31/12/2018.

The investigators will collect all clinical (diagnosis of gout CCPD or hydroxyapatitis, tender and swollen joint count), biological (blood results: ESR, CRP, uric acid, synovial analysis), radiological data (X-rays performed and their description) .

ELIGIBILITY:
Inclusion Criteria:

* Crystal- induced arthritis
* Treatment by biologic
* In western France

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Crystal- induced arthritis Treated by biologic
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Treatment duration | one year
  Duration of treatment by biologic in days

SECONDARY OUTCOMES:
number of synovitis | inclusion
  number of synovitis on 44

CONTACTS AND LOCATIONS:
Overall Officials: Alain SARAUX, MD, PhD, Principal Investigator — CHU Brest
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Undecided